CLINICAL TRIAL: NCT01461083
Title: Phase I Evaluation of [18F]MPPF as a Brain Tracer of Serotonin Receptor 5HT1a in Subjects With Parkinson Disease and Healthy Subjects
Brief Title: Evaluation of [18F]MPPF as a Brain Tracer of Serotonin Receptor 5HT1a
Acronym: MPPF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, David Russell, MD, PhD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MPPF
Record Dates: First submitted 2011-09-27; First posted 2011-10-27 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; [18F]MPPF
MeSH Terms: conditions — Parkinson Disease | interventions — 4-(2'-methoxyphenyl)-1-(2'-(N-2'-pyridinyl)-p-(18F)fluorobenzamido )ethylpiperazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Assess [18F]MPPF and PET imaging (Experimental): To assess [18F]MPPF and PET imaging
  Interventions: Drug: [18F]MPPF

INTERVENTIONS:
Drug: [18F]MPPF — Subjects will be dosed by intravenous bolus injection of [18F]MPPF targeted to be 5.0 mCi, and not to exceed 5.5 mCi (not >10% of 5.0 mCi limit) and not to exceed 5 µg of MPPF

SUMMARY:
The underlying goal of this study is to assess [18F]MPPF PET imaging as a tool to evaluate the activity of the serotonin 5HT1a receptor in the brain of Parkinson Disease (PD) research participants.

DETAILED DESCRIPTION:
Approximately 40 subjects with Parkinson disease and 20 healthy control subjects will be recruited to participate in the 2 Projects in this study. All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations.

Subjects in Project 1 (20 PD and 20 HC subjects) will be asked to undergo a single bolus injection of [18F]MPPF followed by serial Positron Emission Tomography (PET) imaging scans and blood sampling for measurement of [18F]MPPF in plasma (both protein bound and free) over a period of up to 2 hours. The imaging analyses will be performed by an image-processing specialist who will remain masked to the procedures employed with each imaging acquisition. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, [18F]MPPF. Time to the peak uptake and amplitude of the peak uptake will be evaluated for all brain regions and the results for the PD subjects will be compared with the HC subjects.

Subjects participating in Project 2 (20 PD subjects on dopaminergic replacement therapy) will also undergo a second [18F]MPPF and PET imaging session, identical except that PD medications will be withheld for approximately 8 hours prior to the imaging session. The second session will occur greater than 7 days, but not more than 3 months, from the first imaging session. Initial 'on' medication quantitative outcomes for each brain region will be compared to the outcomes from the second 'off' medication imaging session to determine the influence of dopaminergic treatment on 5HT1A activity.

The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, [18F]MPPF. Time to the peak uptake and amplitude of the peak uptake will be evaluated for all brain regions and the results for the PD subjects will be compared with the HC subjects.

ELIGIBILITY:
PD Subjects

Inclusion Criteria:

* The participant is 30 years or older.
* Written informed consent is obtained.
* Participants have a diagnosis of PD (based on UK Brain Bank Criteria).
* Modified Hoehn and Yahr stage of 1 - 4.
* For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F] CFPyPB injection.

Exclusion Criteria:

* The subject has a clinically significant laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Evidence of a stroke or mass lesion in a clinically relevant area that may interfere with the imaging outcome measure
* Subject treated with medication known to interfere with [18F]MPPF binding in vivo (e.g. pindolol)
* Subjects with radiation exposure above acceptable levels, i.e. a history of exposure to any radiation >15 mSv over the past 12 months.

Healthy control subjects

Inclusion criteria:

* The participant is 18 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* For females, non-child bearing potential a negative urine or blood pregnancy test on day of [18F]MPPF injection.

Exclusion criteria:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* Evidence of a stroke or mass lesion in a clinically relevant area that may interfere with the imaging outcome measure
* Subject treated with medication known to interfere with [18F]MPPF binding in vivo (e.g. pindolol)
* Subjects with radiation exposure above acceptable levels, i.e. a history of exposure to any radiation >15 mSv over the past 12 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To assess the dynamic uptake and washout of [18F]MPPF in brain using positron emission tomography(PET) imaging | 2 years
  To assess the dynamic uptake and washout of [18F]MPPF in brain using positron emission tomography (PET) in Parkinson disease and similarly aged healthy control subjects as a potential imaging biomarker of the serotonin (5HT1A) receptor in brain.

SECONDARY OUTCOMES:
To assess the influence of dopaminergic replacement therapy on 5HT1A activity in PD subjects | 2 years
  To assess the influence of dopaminergic replacement therapy on 5HT1A activity in PD subjects

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, MD, PhD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

REFERENCES:
- See also: Institute for Neurodegenerative Disorders — http://www.indd.org